CLINICAL TRIAL: NCT00800761
Title: Increased Survival and Reversion of Iron-Induced Cardiac Disease in Patients With Thalassemia Major Receiving Intensive Combined Chelation Therapy
Brief Title: Intensive Combined Chelation Therapy for Iron-Induced Cardiac Disease in Patients With Thalassemia Major
Acronym: DFODFPTM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Microcitemico (Other)
Collaborators: Azienda Sanitaria Locale di Cagliari (Other)
Responsible Party: Maria Eliana Lai, Prof, MD, Adult Thalassemic Center, Director, University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFO-DFP in TM; DFOplusDFPLAI
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2001-12

CONDITIONS: Iron Overload; Cardiomyopathy
MeSH Terms: conditions — Iron Overload; Cardiomyopathies | interventions — Deferoxamine; Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deferoxamine alone (Active Comparator): comparison of deferoxamine subcutaneous 40mg/kg/die alone versus combined therapy deferoxamine-deferiprone
  Interventions: Drug: Deferoxamine and Deferiprone; Drug: Deferoxamine
- Deferoxamine plus Deferiprone (Active Comparator): comparison of two arms: the first one treated with deferoxamine subcutaneous vials,40 mg/kg,12 hours/die plus deferiprone tablets 75 mg/kg three times/die versus the second one treated with deferoxamine subcutaneous vials,40 mg/kg,12 hours/die
  Interventions: Drug: Deferoxamine and Deferiprone

INTERVENTIONS:
Drug: Deferoxamine and Deferiprone — comparison of two arms: the first one treated with deferoxamine subcutaneous vials,40 mg/kg,12 hours/die plus deferiprone tablets 75 mg/kg three times/die versus the second one treated with deferoxamine subcutaneous vials,40 mg/kg,12 hours/die
Drug: Deferoxamine — deferoxamine vials,40 mg/kg,12 hours/die
  Arms: Deferoxamine alone

SUMMARY:
Myocardial iron overload is the leading cause of death in patients with beta-thalassemia major (TM). Therapy with deferoxamine (DFO) combined with deferiprone (DFP) reduces myocardial iron and improves cardiac function. However, the prognosis for TM patients with established cardiac disease switched from DFO monotherapy to combined DFP/DFO chelation is unknown. Twenty-eight TM patients with cardiac disease were enrolled in a prospective study lasting 42±6 months. Fifteen (9 high-ferritin and 6 low-ferritin) were placed on DFP/DFO (DFP, 75 mg/kg t.i.d.; DFO, 40-50 mg/kg over 8-12 h at night 5-7 d/wk), while 13 (5 high- and 8 low-ferritin) received DFO alone. No cardiac events were observed among high-ferritin patients on combination therapy, whereas 4 cardiac events (p=0.0049), including three deaths, occurred in high-ferritin patients on DFO monotherapy. These findings demonstrate that in TM patients with well-established cardiac disease combined iron-chelation therapy with DFP/DFO is superior to DFO monotherapy.

ELIGIBILITY:
Inclusion Criteria:

Cardiomyopathy secondary to iron overload

Exclusion Criteria:

Heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-12; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Our primary objective: to assess the prevalence of cardiovascular deaths and hospitalisations for cardiovascular disease in the 2 treatment groups | 42 months

SECONDARY OUTCOMES:
monitor the left ventricular ejection fraction (LVEF) and serum ferritin levels for evidence of improvement. | 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Lai, MD, Study Director — Department of Internal Medicine, University of Cagliari-Italy
Locations (1):
- Adult Talassemic Center, Ospedale Microcitemico, Cagliari, Sardinia, Italy

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597